PRINCIPAL INVESTIGATOR: Jonathan M. Hernandez, MD

STUDY TITLE: Perioperative MVT-5873, a Fully Human Monoclonal

Antibody Against a CA 19-9 Epitope, for Operable CA

19-9 Producing Pancreatic Cancers,

Cholangiocarcinomas, and Metastatic Colorectal Cancers

STUDY SITE: NIH Clinical Center

Cohort: Affected Patients

Consent Version: 08/10/2020

### WHO DO YOU CONTACT ABOUT THIS STUDY?

Jonathan M. Hernandez, MD, by phone at 240-760-6072 or email at jonathan.hernandez@nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

In this study we will investigate safety of using MVT-5873 given at the time of surgery to remove your cancer and whether MVT-5873 can increase the time it takes for your disease to get worse.

MVT-5873 is an investigational (has not been approved by the FDA) agent. This is the first study in which the MVT-5873 is being given to humans prior to and after surgery.

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Version Date: 08/10/2020


One of the features of tumors of the gastrointestinal tract is the presence of a molecule called CA 19-9 in the tumors and in the blood. MVT-5873 was designed to target and block CA 19-9. We believe that MVT-5873 can be more effective in patients with CA 19-9 positive tumors, but we do not know for sure. Considering this, we will enroll people with specific level of CA 19-9 in patients' blood.

This study has two parts: safety and efficacy.

First, we are going to evaluate the safety of using MVT-5873 prior to and after surgery to remove your tumor. Increasing doses of MVT-5873 will be given to participants in the study to find the highest dose of MVT-5873 that people can tolerate when given at the time of surgery.

Secondly, we will study if the recommended dose of MVT-5873 at the time of surgery can increase the time it takes for your disease to get worse.

### WHY ARE YOU BEING ASKED TO TAKE PART IN THIS STUDY?

You are being asked to take part in this study because you have been diagnosed with pancreatic cancer, bile duct cancer or colorectal cancer with metastases to the liver, and you have a certain level of CA 19-9 in your blood.

### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Up to 105 people will be enrolled on the study, but because not everyone will be eligible, it is expected that about 83 will be treated.

## **DESCRIPTION OF RESEARCH STUDY**

## Before you begin the study

Before you begin this study, you will need to have the following exams and tests to make sure you are eligible for this study. These exams and tests are part of regular cancer care. If you recently had some of the tests, they may not need to be repeated. You will be removed from the study if you are not eligible:

- A review of any past or current medical conditions, demographic data (your sex, age, race/ethnicity), medicines you have been taking, cancer and its treatment history.
- Physical examination, including height, weight and vital signs.
- Electrocardiogram (EKG a record of your heartbeat) to evaluate your heart.
- Review of your symptoms and your ability to perform your normal activities.
- Imaging Assessments a computed tomographic scan (CT) that produces a picture of your body using a small amount of radiation or magnetic resonance imaging (MRI) that uses a magnetic field to produce an image of your body. These will be used to examine your chest, abdomen, and pelvis.
- Routine blood tests:
  - Tests to find out if you are anemic, have low blood counts, your blood is clotting normally and if your liver, kidneys, and other organs are working well.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- To look at the CA 19-9 level in your blood.
- o Tests for Hepatitis B and C. If you are infected with Hepatitis B or C you will not be able to participate in this study as it will pose additional risk to you. We will tell you what the results mean, how to find care, how to avoid infecting others, and the importance of informing your partners at possible risk because of your infection.
- Serum or urine pregnancy test if you are a woman who can have children.
- You will be asked to provide confirmation of your diagnosis. If tumor sample from a
  previous surgery/biopsy is not available, we will perform a biopsy (collect a sample of your
  tumor) to confirm your diagnosis.

You will also be asked to co-enroll on the Surgical Oncology Program's tissue collection protocol 13C0176 ("Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors") so that any remaining tumor or blood samples that were collected as a part of this study can be used for future research when this study ends.

# **During the Study**

During the study MVT-5873 treatment MVT-5873 will be administered to you through an IV (intravenous catheter, a small plastic tube that is put into a vein, usually in your arm) before and after surgery.

The first infusion will be done 3 to 7 days before surgery (Day -3). This infusion will last approximately 2 hours. If tolerated, the infusion time for subsequent infusions may be shortened.

After your recover from surgery (approximately 1 to 2 weeks after the operation) we will continue administration of MVT-5873 on a 3-week (21 day) cycle basis. During the first 21-day cycle, two infusions will be given a week apart on Day 1 and Day 8, and then every 2 weeks during Cycle 2.

### Surgery

In this study you will be admitted to the hospital for surgery. Most patients are admitted the evening before their operation. Your physician will explain the surgical procedure and will answer any questions you may have. You will be asked to sign a separate consent for the operation.

You will undergo a major surgical operation to remove as many of your visible cancer tumors as possible.

# Recovery

After the operation, you will be admitted to the Intensive Care Unit (ICU) where you will be monitored closely for 1-4 days. As with any major operation, you may have a breathing tube and be connected to a breathing machine for 1-2 days following the operation. You will have a tube in your stomach, a catheter (tube) in your bladder and several IVs during this period. As soon as you are able, you will be helped to get out of bed, to cough and take deep breaths and to walk. Once your bowel function has returned to normal, you will be allowed to eat – this usually takes 5-7 days.

When your condition is stable, you will be transferred to the regular patient care unit until you are ready to be discharged to home, usually 7-14 days following the operation. Throughout your

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


hospitalization, you will receive pain medications, IV fluids, antibiotics, and blood transfusions as necessary.

# **Ongoing Procedures**

While you are on the treatment, every time you visit the Clinical Center for MVT-5873 infusion and surgery, you will have:

- Review of current medical conditions and medicines you are taking.
- Physical examination, including weight and vital signs.
- Review of your symptoms and your ability to perform your normal activities.
- Routine blood tests to find out if you are anemic, have low blood counts, your blood is clotting normally and if your liver, kidneys, and other organs are working well.

During these visits you will also have the following done for research purposes and to check if the treatment is working:

- Research blood tests to look at the CA 19-9 level in your blood. (You will have your CA 19-9 level collected before the study drug infusion and 2 hours after the study drug infusion.)
- Imaging Assessments a computed tomographic scan (CT) that produces a picture of your body using a small amount of radiation or magnetic resonance imaging (MRI) that uses a magnetic field to produce an image of your body. These will be used to examine your chest, abdomen, pelvis.

### Research Tests

In addition to the tests that we will conduct to determine whether you are having side effects or if you are responding to the study therapy, we will also collect samples from you for purposes of research only. Some of the analyses will be done outside of the NIH, but your samples will not contain any information that can identify you.

These studies include:

- Collection of blood before treatment, on day of surgery, on Day 1 of Cycle 1, and at the end of treatment visit to:
  - Measure the amount of tumor cells in your blood, and study how these tumor cells respond to the study therapy.
- During surgery, we will collect tissue samples of your tumor and normal liver to study:
  - How efficiently your genes are working, the difference in proteins, metabolism and microenvironment in your tumor compare to normal tissue.
  - o The long-term effect of treatment on proteins, metabolism and microenvironment in your tumor and normal liver tissue. Your liver tissue will be used in the development of a "liver model" and your samples will be kept "live" in a special device.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


O The molecular mechanisms of tumor development, growth, and response to treatment. We will keep your samples "live" for a short period of time (up to 4 days) and use these samples in the development "SMART System models" - which can test multiple treatments and allow us to study the effect of each treatment and how the treatments compare to each other.

## Genetic testing and return of results

Your tissue samples contain genes, which are made up of DNA (deoxyribonucleic acid) and transcript of these genes made of RNA (ribonucleic acid) which serves as the "instruction book" for the cells that make up our bodies. We will use the tissue samples you provided to learn about how the genes in your tumor compare to genes in normal tissue. Your tissue will help us study how genes might play a role in colon cancer and other diseases. We will not share the results of these research tests with you.

When we are conducting the above genetic tests, it is possible that we could identify changes in other parts of your RNA that are not related to this research. These are known as "incidental medical findings":

- Changes in genes that are related to diseases other than cancer.
- Changes in genes that are not known to cause any disease. These are known as normal variations.
- Changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

However, the analyses that we perform in our laboratory are for research purposes only; they are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing. Changes that we observe unrelated to our research may or may not be valid. Therefore, we do not plan to inform you of the results of testing on your tissue and blood that is performed in our research lab. However, in the unlikely event that we discover a finding that is believed to be clinically important based on medical standards at the time that we first analyze your results, we will contact you. This could be many years in the future. We will ask you to have an additional tube of blood drawn to verify the findings we have seen in our lab. If the results are verified, you will be re-contacted and offered a genetic counseling here at Clinical Center (no charge) or referral to an outside genetic healthcare provider (at your expense) to discuss the results.

# When you are finished taking the drug (treatment)

After completion of the therapy, you will be invited for follow up visits approximately 1 week (end of treatment) and 1 month after the last day you take the study drug. At these visits, you will have the following tests:

- Review of current medical conditions and medicines you are taking.
- Physical examination, including weight and vital signs.
- Review of your symptoms and your ability to perform your normal activities.
- Routine blood tests:

# PATIENT IDENTIFICATION | Consent to Participate in a Clinical Research Study

WILL 2077 (4.17)

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- o Tests to find out if you are anemic, have low blood counts, your blood is clotting normally and if your liver, kidneys, and other organs are working well.
- Imaging Assessments a computed tomographic scan (CT) that produces a picture of your body using a small amount of radiation or magnetic resonance imaging (MRI) that uses a magnetic field to produce an image of your body. These will be used to examine your chest, abdomen, pelvis (only at 1-week visit).

During these visits you will also have the following tests for research purposes:

• Research blood tests to look at the CA 19-9 level in your blood. (This will also be done during your long term follow up.)

If you are not able to come to these visits, we may be able to call/videocall you and arrange for you to have a visit with a home physician, with certain tests done at outside labs nearer to your home and the results sent to us instead. Your healthcare team will let you know more if this is the case. We will contact you by telephone/videocall or email to ask if you have side effects.

After that, we will contact you by telephone/videocall or email every four months to determine your health status and to find out about any new cancer treatments that you have begun. This will continue for the rest of your life or until the study is stopped.

# BIRTH CONTROL, RISKS OF PREGNANCY AND BREASTFEEDING

There may be a high risk that the study treatment may damage an unborn child (embryo or fetus); therefore, if you are a female, you must not get pregnant while in this study. This is why the study doctor will ask if you are using an acceptable method of birth control (contraception) and why you should inform your doctor if you think you may be pregnant.

The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control listed below while in this study (and for 3 months after your last dose). If you become pregnant during the study, you will be discontinued from the study, and your physician will need to follow up with your pregnancy and your child's health.

Acceptable methods of birth control for this study include:

- Norplant
- Birth control pills plus another method (i.e. condom)
- Birth control patch
- IUD (intrauterine device)
- Depo-Provera
- Sterilization
- Abstinence
- Condoms with spermicide

If you are a woman of childbearing age, you must use birth control for the entire duration of the study treatment and for 3 months afterwards or you cannot be in the study. Hormonal methods

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


(birth control pill, etc.), double-barrier methods (condoms with spermicidal, sponge with spermicidal, or diaphragm with spermicidal), or abstinence may be used. Your doctor will discuss these with you. Some methods of birth control will not work when you are taking certain drugs. Be aware that you can still become pregnant even if you use an acceptable birth control method.

The study doctor will require some women who join the study to have pregnancy tests before the study. A pregnancy test does not keep you from becoming pregnant.

If you are a man, there may be risks to an unborn baby you father during or after the study; therefore, you must use birth control if you choose to have sex with women during the study treatment (and for 3 months after your last dose). You must also not donate sperm during the study treatment and for at least 3 months after completion of the study. If you are a male with a partner who could become pregnant, you must use condoms and make sure your partner is also using effective birth control during the study. If your partner becomes pregnant, you must tell the study doctor immediately.

If you think you are or your partner is pregnant during the study, you must tell the study doctor immediately. If you become pregnant, you will have to stop the study treatment. The study doctor may ask for information about the pregnancy and the birth of the baby. The study doctor may share this information with the sponsor and the IRB (organization overseeing the study).

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, the drug or procedure may involve risks to the unborn baby, which are currently unforeseeable.

A pregnancy test can be wrong. If you become pregnant during the study, call the study doctor at once. You will not receive any further treatments with the study drug.

You cannot be in the study if you are pregnant or breastfeeding. It is not known whether the study drug is safe for breast-fed babies. Therefore, if you are breastfeeding a child, then you must stop breastfeeding.

### RISKS OR DISCOMFORTS OF PARTICIPATION

If you do not understand what any of these side effects mean, please ask the study doctor or study staff to explain these terms to you.

Because the study drug is investigational, all of its side effects may not be known. There may be rare and unknown side effects, some of which may be irreversible and/or life-threatening. You should report all side effects that you experience to the study doctor.

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. However, doctors do not know all the side effects that may happen. Side effects may be mild or very serious. The study doctor may give you medicines to help lessen side effects.

You must tell the study doctor or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

If you choose to take part in this study, there is a risk that:

• There may be complications that preclude a surgery with a chance of cure.

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- There may be complications that preclude a treatment with known survival benefit.
- Based on the observation of liver toxicity in prior studies:
  - o The removal of your tumor may be delayed.
  - o The start of chemotherapy after your operation may be delayed.
- A delay in the start of standard adjuvant chemotherapy may affect your outcome.
- You may lose time at work or home.
- You may spend more time in the hospital or doctor's office than usual.
- You may be asked sensitive questions that you normally do not discuss.

The drugs used in this study may affect how different parts of your body work, such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.
- There might be other side effects that researchers do not yet know about. If important new side effects are found in other patients participating in this study, the study doctor will discuss these with you.

#### **MVT-5873**

To date, forty-nine (49) patients have received the study drug MVT-5873. All possible side effects of the study drug are not yet known. In this limited number of patients, the study drug has been known to cause side effects typically seen with other antibodies. The side effects have gone away after the study drug is stopped, but some side effects could be serious and long lasting.

- Allergic reactions, consisting of one or more of the following:
  - Fever
  - o Chills

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- o Nausea
- Vomiting
- Headache
- o Rashes, including hives
- Dizziness
- Difficulty breathing
- Shortness of breath
- Wheezing
- Chest tightness
- Lowered blood pressure
- Diarrhea or loose stools
- Fatigue
- Fever
- Increase in blood levels that measure liver function
- Pneumonitis (inflammation of the lung wall) was observed in some patients receiving MVT-5873 in combination with the gemcitabine plus nab-paclitaxel chemotherapy

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

When you take more than one drug at a time, the side effects can be worse or different than if you take either drug by itself.

Until you know how the study drug will affect you, you should use caution by avoiding stairs, not driving a car or working with machinery.

You may form antibodies to the drug. An antibody is a type of protein that helps protect the body against attack by bacteria and viruses. There is also a small chance that if you have these antibodies, this drug or similar drugs will not work for you in the future.

Please tell the study doctor or study staff right away if you have any side effects. Please tell them if you have any other problems with your health or the way you feel during the study, regardless of whether or not you think these problems are related to the investigational drug.

# Could I have an allergic reaction?

Sometimes people have allergic reactions to drugs. If you have a very bad allergic reaction, you could die. Some things that happen during an allergic reaction are:

- A rash
- Having a hard time breathing
- Wheezing

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY
- A sudden drop in blood pressure (making you feel dizzy or lightheaded)
- Swelling around the mouth, throat or eyes
- A fast pulse
- Sweating

You should get medical help and contact the study doctor or study staff if you have any of these or any other side effects during the study.

# Could I have any other problems with my health if I do this research study?

It is possible that receiving this study drug with your regular medications or supplements may change how the study drug, your regular medications, or your regular supplements work. It is very important that you tell the study doctor about all medications or supplements you are taking during the study.

### ADDITIONAL RISKS OR DISCOMFORTS

# **Blood Samples**

There may be side effects of having blood drawn taken by single needle-sticks or by a tube that is left in your arm such as:

- Fainting
- Redness
- Pain
- Bruising
- Bleeding
- Infection
- Blood clots, which may cause inflammation, swelling and pain

If you feel faint tell the study staff right away.

# Risks of using an Intravenous (IV) Catheter

- Infection
- Pain
- Redness
- Bruising
- Vein irritation from the fluids or medication being given
- Local swelling due to IV fluid accidentally entering the tissue rather than the vein
- Blood clots, which may cause inflammation, swelling and pain

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


### **Tissue Collection Risk**

We will use some of the tissue we collect from your liver during your standard of care surgery for research. If you do not need to remove a part of your liver as part of your treatment, we will take a small sample from your liver for research purposes during the standard of care surgery on your pancreas. There is a slight risk this may cause additional bleeding, infection or damage to your liver.

# **Risks from Biopsy**

This procedure usually causes only brief discomfort at the site from which the biopsy is taken. Rarely, infection or bleeding may occur at the needle site. Tumor biopsy will be done by a specialist using the CT scanner or ultrasound to guide the biopsy needle into the tumor to ensure accuracy. We will give you more information about the risks of radiation during the CT guided biopsies on this study in this consent form below.

# **Surgery**

The risks of undergoing a resection will be specific to your operation. Dr. Hernandez will discuss the specific risks in detail during the procedural consent, which will be obtained separately from the study consent in accordance with NIH policy.

#### **Urine Collection**

There is no physical risk involved with urine collection.

## Electrocardiogram (EKG)

This test evaluates your heart rate and rhythm by measuring electrical impulses from the heart through electrodes that are placed on the skin. You must lie down and be still without talking during the 5 minutes the EKG is being recorded. This procedure is associated with minimal discomfort.

#### **Scans and Contrast**

CT and MRI scans are common standard imaging tests used in the diagnosis of cancer. The most common discomfort is the length of time a patient must lay still during a scan. Occasionally, a patient may become uncomfortable with the closed space of the machines, particularly the MRI. If this occurs, your doctor can order a medicine to help you relax during this scan. If a contrast agent (the special dye) is given with the scan there is a small risk of having a reaction to the contrast. In that small group of patients who have a reaction, the most common symptoms are nausea, pain in the vein where the contrast was given, a metallic or bitter taste in the mouth, and a warm or flushing feeling that lasts from 1-3 minutes. Rarely do these symptoms require any treatment. In very rare cases, people have had severe reactions that affect their breathing and heart rhythm. If you have had a reaction in the past, be sure to tell you doctor or nurse about it.

An IV line may need to be inserted for administration of the contrast agent or anesthetic. This can cause pain at the site where the IV is placed and carries a small risk of bruising or infection.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis" which has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is not normal or if you received gadolinium within the previous month.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA recently issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain, whenever possible. We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

Patients with a cardiac pacemaker, neural pacemaker, some types of surgical clips, cochlear implants, foreign metal objects, permanent retainers, or any iron-containing material within the body should not undergo MRI, because of the effect of the strong magnet on these objects.

# What are the risks of radiation from being in the study?

During your participation in this research study, you will be exposed to radiation from CT scans. The amount of radiation exposure you will receive from these procedures is equal to approximately 8.5 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." This study will expose you to more radiation than you get from everyday background radiation. No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT scans that you get in this study will expose you to the roughly the same amount of radiation as 28.3 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 0.9 out of 100 (0.9%) and of getting a fatal cancer is 0.4 out of 100 (0.4%).

### Psychological or Social Risks Associated with Return of Incidental or Secondary Findings

As part of the research study, it is possible that you could learn that you have genetic risks for another disease or disability. This may be upsetting and, depending on what you learn, might create a need to make challenging decisions about how to respond.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


Although your genomic information is unique to you, you share some genomic similarities with your children, parents, brothers, sisters, and other blood relatives. Therefore, learning your research results could mean something about your family members and might cause you or your family distress. Before joining the study, it may be beneficial to talk with your family members about whether and how they want you to share your results with them.

# Privacy Risks Associated with Return of Incidental or Secondary Findings

Although your genetic information is unique to you, you do share some genetic information with your children, parents, brothers, sisters, and other blood relatives. Consequently, it may be possible that genetic information from them could be used to help identify you. Similarly, it may be possible that genetic information from you could be used to help identify them. Patterns of genetic variation also can be used by law enforcement agencies to identify a person or his/her blood relatives.

## **Protections Against Misuse of Genetic Information**

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

#### POTENTIAL BENEFITS OF PARTICIPATION

# Are there benefits to taking part in this study?

The aim of this study is to see if this experimental treatment will make persons with your disease live longer. We do not know if you will receive personal, medical benefit from taking part in this study. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the treatment's effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer

### ALTERNATIVE APPROACHES OR TREATMENTS

### What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options:

- Getting treatment or care for your cancer without being in a study.
- Taking part in another study.
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


Please talk to your doctor about these and other options.

#### STOPPING THERAPY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease gets worse during treatment
- if you develop unacceptable toxicity to study treatment
- if you need chemotherapy
- if you become pregnant
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases can**not** be recalled and destroyed.

### CONFLICT OF INTEREST

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest

### USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

Your samples will be stored for future use under the seperate specimen collection protocol (13C0176) in which you have agreed to be co-enrolled.

To advance science, it is helpful for researchers to share information they get from studying human data. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use data stored in scientific databases to advance science and learn about health and disease.

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


We plan to keep some of your specimens and data that we collect on this study and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared with be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

# **Genomic Data Sharing**

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity, and sex. If your individual data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

Summary information about all of the participants included in this study (including you) is being placed in a database and will be available through open access. That means that researchers and non-researchers will be able to access summary information about all the participants included in the study, or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you with this information is very low.

NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

## COMPENSATION, REIMBURSEMENT, AND PAYMENT

### Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


The NCI generally does not cover expenses during screening. If you are scheduled for and begin treatment, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. Someone will work with you to provide more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- Qualified representatives from AAIPharma, the pharmaceutical company who produces MVT-5873.

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens or data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)


File in Section 4: Protocol Consent (2)


### **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


## PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Dr. Jonathan Hernandez, MD, jonathan.hernandez@nih.gov, 240-760-6072. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

## **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


IRB NUMBER: 19C0039
IRB APPROVAL DATE: 09/15/2020


| to discuss it and to ask question | | |
|---|---|---|
| Signature of Research Particip | ant Print Name of Research P | articipant Date |
| about this study and have been<br>to make research decisions on | ntative (LAR) for an Adult Unable to Cora given the opportunity to discuss it and to ask behalf of the adult participant unable to consercable, the information in the above consent was to participate in the study. | questions. I am legally authont and have the authority to pro |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | r Date |
| | m consent process only: This section is only English consent form has been approved by t | |
| short-consent process and this translation. | | |
| short-consent process and this translation. Witness: Signature of Witness* *NIH ADMINISTRATIVE INTERPRETER: An interpreter, or other in the administration of informe also serve as the witness. An interpreter, or other in | Print Name of Witness SECTION TO BE COMPLETED RECONDED and the participal dividual, who speaks English and the participal consent and served as a witness. The investigations of the participal consent but did not serve as a witness. The next dividual, who speaks English and the participal consent but did not serve as a witness. The next dividual, who speaks English and the participal consent but did not serve as a witness. The next dividual serves are served as a witness. | Date GARDING THE USE OF ant's preferred language facilitigator obtaining consent may ant's preferred language facilitigator obtaining consent may |

CC ICF template v. 09.27.19